CLINICAL TRIAL: NCT02752529
Title: The Establishment of Multiple Point Prediction Model About Tacrolimus Metabolic Differences Based on Genetic Network After Liver Transplantation and the Application of Multicenter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Peng Zhihai, Director, Head of General Surgery, Principal Investigator, Clinical Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PZhihai
Record Dates: First submitted 2016-03-30; First posted 2016-04-27 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Cirrhosis, Liver
Keywords: Liver Transplantation; Individualized Therapy; Polymorphism
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Tacrolimus/dose1 (Experimental): Tacrolimus 5mg tablet and dosage based on Co once/twice a day for 7 days
  Interventions: Drug: Tacrolimus（FK506）
- Tacrolimus/dose2 (Active Comparator): Tacrolimus 5mg tablet and dosage based on Co once/twice a day for 7 days
  Interventions: Drug: Tacrolimus（FK506）

INTERVENTIONS:
Drug: Tacrolimus（FK506）

SUMMARY:
Combined with the clinical data of FK506 and the database of GO and Kyoto Encyclopedia of Genes and Genomes（KEGG）, the investigators aim to carry out the bioinformatic analysis and build a muti-locus genetic model, then muti-center assess the predictive accuracy of FK506 metabolic differences.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of end-tage liver diseases
* 18 years old or above
* Han nationality
* Therapeutic regimen：TAC

Exclusion Criteria:

* Less than 18 years old
* Other races
* Therapeutic regimen：cyclosporine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Tacrolimus | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ou B, Liu Y, Zhang T, Sun Y, Chen J, Peng Z. TLR9 rs352139 Genetic Variant Promotes Tacrolimus Elimination in Chinese Liver Transplant Patients During the Early Posttransplantation Period. Pharmacotherapy. 2019 Jan;39(1):67-76. doi: 10.1002/phar.2204. Epub 2019 Jan 8. PMID 30537010
- [Derived] Zhang T, Liu Y, Zeng R, Ling Q, Wen P, Fan J, Peng Z. Association of donor small ubiquitin-like modifier 4 rs237025 genetic variant with tacrolimus elimination in the early period after liver transplantation. Liver Int. 2018 Apr;38(4):724-732. doi: 10.1111/liv.13597. Epub 2017 Oct 4. PMID 28941036